CLINICAL TRIAL: NCT06558994
Title: Transection Versus Ligation of Internal Spermatic Vessels in First Stage Laparoscopic Fowler-Stephens Orchidopexy for Intra-abdominal Testis. Randomized Study
Brief Title: Transection Versus Ligation of Internal Spermatic Vessels in Laparoscopic Fowler-Stephens Orchidopexy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Mohamed Atef Abdelaziz Mostafa, Lecturer of Urology, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ahmed Hassan Protocol
Record Dates: First submitted 2024-08-12; First posted 2024-08-19 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Cryptorchidism
MeSH Terms: conditions — Cryptorchidism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transection arm (Active Comparator): Transection of internal spermatic vessels in first stage laparoscopic Fowler-Stephens orchidopexy for intra-abdominal testis
  Interventions: Procedure: Transection of internal spermatic vessels in first stage laparoscopic Fowler-Stephens orchidopexy for intra-abdominal testis
- Ligation arm (Active Comparator): ligation of internal spermatic vessels in first stage laparoscopic Fowler-Stephens orchidopexy for intra-abdominal testis
  Interventions: Procedure: Ligation of internal spermatic vessels in first stage laparoscopic Fowler-Stephens orchidopexy for intra-abdominal testis

INTERVENTIONS:
Procedure: Transection of internal spermatic vessels in first stage laparoscopic Fowler-Stephens orchidopexy for intra-abdominal testis — Half of the patients will undergo transection of internal spermatic vessels in first stage laparoscopic Fowler-Stephens orchidopexy for intra-abdominal testis.
  Arms: Transection arm
Procedure: Ligation of internal spermatic vessels in first stage laparoscopic Fowler-Stephens orchidopexy for intra-abdominal testis — Half of the patients will undergo ligation of internal spermatic vessels in first stage laparoscopic Fowler-Stephens orchidopexy for intra-abdominal testis
  Arms: Ligation arm

SUMMARY:
This is a comparative study to see the outcome of yransection versus ligation of internal spermatic vessels in first stage laparoscopic Fowler-Stephens orchidopexy for intra-abdominal testis in assisting the descent of the testis to the base of scrotum during the second stage

DETAILED DESCRIPTION:
Cryptorchidism is one of the most commin congenital deformities of male newborns, known as undescended testis (UDT). The incidence ranges according to gestational age, affecting 1.0-4.6% of full-term infants and 1.1-45% of preterm infants. (UDT) is a condition in which the testicles are not found at the base of the scrotum. Studies have shown that the undescended testicle has a potential of spontaneous descent during the first 3 months of life and is less likely to do so after 6 months of age. In almost 20% of cases the undescended testes are not palpable, increasing the difficulty of investigations and treatment, and 30% of these cases are also intra-abdominal. If UDT left untreated, it can cause histological alterations of the testicular cells and increasing of the risks of infertility.

As of treatment of UDT, laparoscopic surgery is ,for most surgeons, the preferred technique. Several techniques have been described for laparoscopic orchidopexy. After spermatic vascular transection, single-stage testicular descent fixing was carried out, as Fowler and Stephens (FSO) first described in 1959. Since 1996, a two-stage laparoscopic Fowler-Stephens technique involving preservation of the gubernacular vessels and performing an entirely laparoscopic second stage. The second stage is presently performed 6-9 months after the first.

Recently, laparoscopic FSO has been adopted to treat high-level IATs, for its minimally invasive wound and acceptable success rate.

ELIGIBILITY:
Inclusion Criteria:

All patients with Unilateral or Bilateral impalpable testis

Exclusion Criteria:

1. Previous Laparotomy surgery
2. Previous Ventriculo-peritoneal shunt
3. Previous laparoscopy for impalpable testis (outside study)
4. Previous Inguinal/Scrotal surgery
5. Disorder of sexual differentiation
6. Abnormal Karyotyping
7. Intra-operative Inguinal testis
8. Ipsilateral testis : Peeping/ Vas internal internal ring / Vanished / Streak / Ovotestis / Ovary.
9. Contralateral : Streak/ Ovotestis/ Ovary

Max Age: 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 58 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
testis-to-ring distance in mm at the second stage | At 6 months after the first stage (during the second stage)
  After either of transection or ligation of the spermatic vessels during the first stage of laparoscopic Fowler-Stephens orchidopexy, the location of the testis away from the internal inguinal ring (the testis-to-ring distance in mm) will be measured during the 2nd stage (degree of descent) 6 months after the first stage and compared among the two groups.
Testicular volume in mL | At 6 months after the first stage (during the second stage)
  After either of transection or ligation of the spermatic vessels during the first stage of laparoscopic Fowler-Stephens orchidopexy, the testicular volume in mL will be assessed intraoperatively during the second stage (6 months after the first stage) and compared among the two groups.

SECONDARY OUTCOMES:
Operative time in minutes | At 6 months after the first stage (during the second stage)
  After either of transection or ligation of the spermatic vessels during the first stage of laparoscopic Fowler-Stephens orchidopexy, the operative time in minutes of the second stage will be measured and compared among the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa M. Mostafa, MD, MSc, PhD, Principal Investigator — Assiut University
Locations (1):
- Assiut University Urology Hospital, Asyut, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be made available to protect privacy of patients

REFERENCES:
- [Background] Virtanen HE, Bjerknes R, Cortes D, Jorgensen N, Rajpert-De Meyts E, Thorsson AV, Thorup J, Main KM. Cryptorchidism: classification, prevalence and long-term consequences. Acta Paediatr. 2007 May;96(5):611-6. doi: 10.1111/j.1651-2227.2007.00241.x. PMID 17462053
- [Background] Vikraman J, Hutson JM, Li R, Thorup J. The undescended testis: Clinical management and scientific advances. Semin Pediatr Surg. 2016 Aug;25(4):241-8. doi: 10.1053/j.sempedsurg.2016.05.007. Epub 2016 May 11. PMID 27521715
- [Background] Wenzler DL, Bloom DA, Park JM. What is the rate of spontaneous testicular descent in infants with cryptorchidism? J Urol. 2004 Feb;171(2 Pt 1):849-51. doi: 10.1097/01.ju.0000106100.21225.d7. PMID 14713841
- [Background] Wang CY, Wang Y, Chen XH, Wei XY, Chen F, Zhong M. Efficacy of single-stage and two-stage Fowler-Stephens laparoscopic orchidopexy in the treatment of intraabdominal high testis. Asian J Surg. 2017 Nov;40(6):490-494. doi: 10.1016/j.asjsur.2016.11.008. Epub 2017 Apr 12. PMID 28410943
- [Background] AbouZeid AA, Mousa MH, Soliman HA, Hamza AF, Hay SA. Intra-abdominal testis: histological alterations and significance of biopsy. J Urol. 2011 Jan;185(1):269-74. doi: 10.1016/j.juro.2010.09.026. PMID 21075394
- [Background] Hvistendahl GM, Poulsen EU. Laparoscopy for the impalpable testes: experience with 80 intra-abdominal testes. J Pediatr Urol. 2009 Oct;5(5):389-92. doi: 10.1016/j.jpurol.2009.04.004. Epub 2009 May 19. PMID 19457721
- [Background] Murphy F, Paran TS, Puri P. Orchidopexy and its impact on fertility. Pediatr Surg Int. 2007 Jul;23(7):625-32. doi: 10.1007/s00383-007-1900-3. Epub 2007 Mar 13. PMID 17431642
- [Background] Chang B, Palmer LS, Franco I. Laparoscopic orchidopexy: a review of a large clinical series. BJU Int. 2001 Apr;87(6):490-3. doi: 10.1046/j.1464-410x.2001.00100.x. PMID 11298040
- [Background] FOWLER R, STEPHENS FD. The role of testicular vascular anatomy in the salvage of high undescended testes. Aust N Z J Surg. 1959 Aug;29:92-106. doi: 10.1111/j.1445-2197.1959.tb03826.x. No abstract available. PMID 13849840
- [Background] Robertson SA, Munro FD, Mackinlay GA. Two-stage Fowler-Stephens orchidopexy preserving the gubernacular vessels and a purely laparoscopic second stage. J Laparoendosc Adv Surg Tech A. 2007 Feb;17(1):101-7. doi: 10.1089/lap.2006.0565. PMID 17362185
- [Background] Humphrey GM, Najmaldin AS, Thomas DF. Laparoscopy in the management of the impalpable undescended testis. Br J Surg. 1998 Jul;85(7):983-5. doi: 10.1046/j.1365-2168.1998.00748.x. PMID 9692579
- [Background] Yu C, Long C, Wei Y, Tang X, Liu B, Shen L, Dong X, Lin T, He D, Wu S, Wei G. Evaluation of Fowler-Stephens orchiopexy for high-level intra-abdominal cryptorchidism: A systematic review and meta-analysis. Int J Surg. 2018 Dec;60:74-87. doi: 10.1016/j.ijsu.2018.10.046. Epub 2018 Nov 5. PMID 30408514